CLINICAL TRIAL: NCT01069770
Title: Neoadjuvant Sunitinib Therapy in Patients With Metastatic Clear Cell Type Renal Cell Carcinoma Patients: a Prospective Study
Brief Title: Neoadjuvant Sunitinib Treatment for Metastatic Clear Cell Renal Cell Carcinoma (RCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Urological Oncology Society (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sung-Goo Chang/ President, Korean Urological Oncology Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sutent-IIR
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastasis
Keywords: Neoadjuvant Therapy; Sunitinib; Clear Cell Renal Cell Carcinoma; Metastasis
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sunitinib — 50mg daily(4 weeks on & 2 weeks off), 2 cycles, until progression or unacceptable toxicity develops
  Other Names: Sutent

SUMMARY:
The purpose of this study is to see whether neoadjuvant administration of Sunitinib reduces the size of the primary kidney tumor in patients with metastatic disease undergoing cytoreductive surgery. The study will also assess the safety of neoadjuvant Sunitinib, objective response rate, respectability of primary tumor, quality of life, and survival advantages.

DETAILED DESCRIPTION:
Primary objectives :

1. Response rate of primary tumor based on RECIST criteria

Secondary objectives :

1. Resectability based on R0 resection rate (negative margin)
2. Toxicities of therapy with neoadjuvant Sunitinib in renal cell carcinoma
3. Quality of life assessed by EORTC QLQ-C30 questionnaire Korean version
4. To assess the efficacy of neoadjuvant therapy of Sunitinib by evaluating time to progression
5. Overall survival rate after Sunitinib therapy
6. Pathologic evaluation after Sunitinib therapy: the change of necrosis and microvessel density

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven RCC with a component of clear cell type histology
* Clinical stage TxNxM+
* At least one site of measurable disease as defined by RECIST criteria
* Potential candidates for cytoreductive nephrectomy
* Favorable or intermittent risk group according to MSKCC risk factor model
* ECOG performance status 0 or 1
* Adequate organ function as defined by:

  * AST or ALT less than or equal to 2.5 times the upper limit of normal
  * Bilirubin less than or equal to 1.5 times the upper limit of normal
  * Absolute neutrophil count (ANC) greater than or equal to 1500/mL
  * Platelets greater than or equal to 100,000/mL
  * Hemoglobin greater than or equal to 9.0 g/dL
  * Serum calcium less than or equal to 12.0 mg/dL
  * Serum creatinine less than or equal to 1.5 times the upper limit of normal
* Male or female, 18 years of age or older
* Women of childbearing potential must NOT be pregnant (as confirmed by a negative pregnancy test)
* Signed informed consent form indicating that the patient or acceptable representative has been informed of all parts of the trial prior to Sunitinib administration (enrollment)
* Willingness and ability to comply with study procedures

Exclusion Criteria:

* History of another primary malignancy within 5 years, with the exception of non-melanoma skin cancer and in situ carcinoma of the uterine cervix.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of commence of Sunitinib therapy.
* Presence of brain metastases during screening period
* Ongoing cardiac dysrhythmias of NCI CTCAE grade of 2 or more, atrial fibrillation of any grade or prolongation of QTc interval to more than 450 millisecond (msec) for male or more than 470 msec for female
* Hypertension that cannot be controlled by medications
* Concurrent treatment with therapeutic doses of coumadin but low dose of coumadin up to 2 mg orally daily for deep vein thrombosis prophylaxis is allowed.
* Current treatment on another therapeutic clinical trial. Supportive care trials or non-treatment trials are allowed.
* Inability to swallow oral medications, or presence of active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea.
* Concurrent medication with known potent CYP3A4 inhibitors and inducers and/or dosing before 7 and 12 days before date of randomization.
* Other severe acute or chronic medical or psychiatric condition of laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Any of the following within 12 months prior to study drug administration:

severe/unstable angina, myocardiac infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.

* Known hypersensitivity to Sunitinib
* Women who are breast-feeding ※ Note At screening, resectability of primary tumor itself does not influence on patients enrollment. Physicians only have to describe about the resectability ("resectable" or "unresectable") at screening on their own discretion, but if they decide that primary tumor is "unresectable", the should specify reasons for unresectable status as follows: invasion into neighboring organs, proximity to vital structure or vessels, bulky regional lymph nodes, vascular invasion, burden of metastatic disease, and others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Response rate of primary tumor based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria | within first 1 week (plus or minus 5 days) after 2 cycles of Sunitinib treatment (1 cycle: 4 weeks on + 2 weeks off)

SECONDARY OUTCOMES:
Overall survival rate after Sunitinib therapy | 2 years
Pathologic evaluation after Sunitinib therapy | After nephrectomy (within 1-6 week after 2 cycles of Sunitinib treatment)
Quality of life (QoL) assessed by EORTC QLQ-C30 questionnaire (Korean version) | 2 years
Resectability based on R0 resection rate | on nephrectomy (within 1-6 week after 2 cycles of Sunitinib treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sungjoon Hong, M.D., Ph.D, Principal Investigator — The Korean Urological Oncology Society
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Seoul
  - Chungbuk University Hospital, Cheonju

REFERENCES:
- See also: Home page of the sponsor's Web site — http://www.kuos.or.kr